CLINICAL TRIAL: NCT02322502
Title: Emergence Times and Airway Reactions in General Laryngeal Mask Airway Anesthesia: a Randomized Multicenter Controlled Trial (ACC Baxter)
Brief Title: Emergence Times and Airway Reactions in General Laryngeal Mask Airway Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-073
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia With Use of LMA (Laryngeal Mask Airway)
Keywords: laryngeal mask airway; desflurane; sevoflurane; propofol
MeSH Terms: interventions — Desflurane; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- desflurane (Experimental): Suprane® Dose: 0.8 MAC / 4-5 vol. % Mode of administration: inhalation with laryngeal mask One application
  Interventions: Drug: Desflurane
- sevoflurane (Active Comparator): Sevoflurane:
  Dose: 0.8 MAC / 1.2-1.4 vol.% Mode of administration: inhalation with laryngeal mask One application
  Interventions: Drug: Sevoflurane
- propofol (Active Comparator): Propofol Dose: 5-7 mg kg-1 h-1 to maintain a BIS index value between 40 and 60 Mode of administration: intravenous One application
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Desflurane — inhalation with laryngeal mask to maintain anaesthesia
  Other Names: Suprane
  Arms: desflurane
Drug: Sevoflurane — inhalation with laryngeal mask to maintain anaesthesia
  Other Names: Sevorane
  Arms: sevoflurane
Drug: propofol — intravenous injection to maintain anaesthesia
  Other Names: Anesia
  Arms: propofol

SUMMARY:
The aim of this study is first to assess if desflurane is superior in order to achieve a faster emergence from anesthesia.

DETAILED DESCRIPTION:
The aim of this study is first to assess if desflurane is superior in order to achieve a faster emergence from anesthesia (stating the date of birth) and second if desflurane is non-inferior in the occurrence of airway complications compared to sevoflurane or total intravenous anesthesia with propofol in the setting of laryngeal mask airway.

ELIGIBILITY:
Inclusion Criteria:

* Planned anesthesia with use of LMA (laryngeal mask airway)
* Planned duration of anesthesia between 0.5 and 2 hours
* Age between 18-75 years
* Both gender
* Body mass index (BMI) <35
* ASA 1-3
* Written informed consent prior to study participation

Exclusion Criteria:

* Planned additional regional and local anesthesia
* Contra-indication for the use of a laryngeal mask airway
* Asthma
* COPD IV
* Known allergy or hypersensitivity to any drugs administered during this study
* Women who are pregnant, breast-feeding or women of childbearing potential not using adequate contraceptive methods
* Participation in a drug or device trial within the previous 30 days.
* Patients legally unable to give written informed consent.
* Patients with severe psychiatric disorders
* Recent (<6 months) history of alcohol or drug abuse
* Patients with severe neuropsychiatric disorders
* Non-fluency in German language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
time of emergence from anesthesia | up to 15 minutes
  time of emergence from anesthesia defined as time between cessation of anesthesia until patient is able to state his/her date of birth on command

SECONDARY OUTCOMES:
Airway reactions (Incidence of intraoperative coughs, laryngospasm) | up to 2 hours
  Incidence of intraoperative coughs (induction/maintenance) - non-inferiority design Incidence of intraoperative laryngospasm (induction/maintenance) Incidence of cough at emergence Incidence of laryngospasms at emergence
Emergence times | up to 15 minutes
  Time to remove laryngeal mask Time to open eyes on command Time to respond on command (press hand) Time to state the name on command Recovery Index (RI = 1 + Aldrete5min/[(2xextubation time) + 1 x opening eyes time)]

CONTACTS AND LOCATIONS:
Overall Officials: Mark Coburn, Prof., Principal Investigator — University Hospital, Aachen
Locations (4):
- Germany (4):
  - RWTH Aachen University; Department of Anesthesia, Aachen
  - Martha-Maria Hospital Halle Dölau gGmbH, Department of Anesthesia, Halle
  - Kreiskliniken Reutlingen, Department of Anesthesia, Reutlingen
  - University Hospital Ulm, Department of Anesthesia, Ulm

REFERENCES:
- [Derived] Kowark A, Rossaint R, Puhringer F, Keszei AP, Fritz H, Froba G, Rex C, Haas H, Otto V, Coburn M; Study Collaborators. Emergence times and airway reactions during general anaesthesia with remifentanil and a laryngeal mask airway: A multicentre randomised controlled trial. Eur J Anaesthesiol. 2018 Aug;35(8):588-597. doi: 10.1097/EJA.0000000000000852. PMID 29916859
- [Derived] Stevanovic A, Rossaint R, Keszei AP, Fritz H, Froba G, Puhringer F, Coburn M. Emergence times and airway reactions in general laryngeal mask airway anesthesia: study protocol for a randomized controlled trial. Trials. 2015 Jul 26;16:316. doi: 10.1186/s13063-015-0855-2. PMID 26210907